CLINICAL TRIAL: NCT03752632
Title: Veinplicity for Improved Venous Access: The VIVA Trial
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business reasons not related to safety or trial conduct
Sponsor: Physeon GmbH (Industry)
Collaborators: Regulatory and Clinical Research Institute Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHY0011
Record Dates: First submitted 2018-11-13; First posted 2018-11-26 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Difficult-to-access Veins for Intravenous Cannulation
Keywords: intravenous; peripheral vein; cannulation; IV access
MeSH Terms: interventions — Tourniquets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Veinplicity with tourniquet (treatment) (Experimental): Veinplicity with tourniquet
  Interventions: Device: Veinplicity with tourniquet
- Tourniquet (control) (Active Comparator): Control: Tourniquet
  Interventions: Device: Tourniquet

INTERVENTIONS:
Device: Veinplicity with tourniquet — Veinplicity will be used with a tourniquet
  Arms: Veinplicity with tourniquet (treatment)
Device: Tourniquet — A tourniquet alone will be used.
  Arms: Tourniquet (control)

SUMMARY:
This study will assess the safety and effectiveness of the Veinplicity device to improve the visualization and palpability of difficult-to-access veins for intravenous cannulation.

DETAILED DESCRIPTION:
This is a prospective, randomized controlled study that will assess ability of Veinplicity to improve successful peripheral vein cannulation at the first stick in enrolled subjects. Potential subjects will undergo a peripheral vein assessment by a study clinician, which is standard of care prior to peripheral vein cannulation (PVC) for the establishment of intravenous (IV) access. Adults who are assessed as having "fair or poor" vein quality will be consented, enrolled and randomized into the study. Subjects will be randomized in a 1:1 ratio to either (1) tourniquet alone (control group); or (2) Veinplicity with tourniquet (treatment group). The primary endpoint is first-stick success. Clinicians will use an 18-, 20- or 22-gauge cannula. Clinician and subject satisfaction will be separately assessed using surveys on Day 0. Subjects in both groups will be followed for one day (either phone or in-hospital visit) after enrollment for safety. Qualified study clinicians must have at least one year of experience inserting peripheral IVs and must perform an average of five PVCs per week. The primary hypothesis to be tested is: Veinplicity with tourniquet is superior to tourniquet alone for successful peripheral vein access at first stick when used to cannulate subjects assessed as having a fair or poor level of vein quality. It is expected that this study will enroll approximately 246 subjects; 123 per study group. It is expected that up to five sites will be involved in this study. A planned interim analysis will be conducted to reassess the study planned sample size when approximately 50% of subjects have been enrolled. Enrollment will not stop during the interim analysis activities. Safety will be evaluated by the collection and analysis of the incidence and severity of all procedure- and/or device-related adverse events through the Day 1 phone call/visit.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 22 years old.
* Subject is assessed as having fair or poor vein quality.
* Subject's both arms are suitable for cannulation.
* Subject will not suffer harm from a delay in having an IV established as determined by the treating clinician.

Exclusion Criteria:

* Subject has existing intravenous access.
* Subject has a planned or existing intra-arterial access.
* Subject has broken, infected or irritated skin and/or dermatological conditions, e.g., eczema, psoriasis and/or allergic reactions, on either forearm.
* Subject has an active implantable medical device.
* Subject wears a transdermal drug delivery patch on her/his forearm.
* Subject has an active/suspected deep vein thrombosis or thrombophlebitis, impaired circulation, impaired sensation, active/uncontrolled bleeding, recently radiated tissue, recent fracture, recent injury or surgery resulting in blood loss > 100 mL, osteoporosis, localized abscess, localized tuberculosis, and/or a chronic wound with potential underlying osteomyelitis.
* Subject has impaired cognition or communication (unable to provide accurate feedback).
* Subject has a history of seizures and/or epilepsy, and/or a recent seizure, possible recent seizure or a history of possible seizures.
* Subject is pregnant and/or breastfeeding at the time of study enrollment.
* Subject has, at the site of or in between Veinplicity electrode application sites, an active/suspected malignancy.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
First-stick success when accessing a peripheral vein for cannulation | Day 0
  successful peripheral vein access for the first-stick with use of Veinplicity with tourniquet versus tourniquet alone
Device and/or procedure-related adverse events | Day 1
  Safety will be evaluated by the collection and analysis of the incidence and severity of all procedure- and/or device-related adverse events through the Day 1 post-insertion phone call/visit.

OTHER OUTCOMES:
Number of attempted sticks to successful vein access | Day 0
  Number of attempted sticks to successful vein access
Total procedure time | Day 0
  For control subjects, timing begins at the start of skin preparation or tourniquet application on the first arm (whichever is first per standard of practice) to either obtaining successful vein access or until the fourth attempt at cannulation fails. For Veinplicity subjects, timing begins at the start of electrode application on the first arm to either obtaining successful vein access or until the fourth attempt at cannulation fails.
Time to first-stick success | Day 0
  time from tourniquet application for the initial cannulation attempt to declaration of first-stick success/failure.
Subject Satisfaction Survey question for control subject's: Past IV starts have been difficult, uncomfortable or painful. | Day 0 after completion of the study procedure
  Control subject's assessment of pain associated with past IV starts:
  Scale 1 - 5; Unable to Evaluate
  1. Strongly Agree
  2. Agree
  3. Neutral
  4. Disagree
  5. Strongly Disagree Unable to Evaluate
Subject Satisfaction Survey question for control subject's: Today, my IV was started easily. | Day 0 after completion of the study procedure
  Control subject's assessment of how easy they believe today's IV start was:
  Scale 1 - 5; Unable to Evaluate
  1. Strongly Agree
  2. Agree
  3. Neutral
  4. Disagree
  5. Strongly Disagree Unable to Evaluate
Subject Satisfaction Survey question for control subject's: Pain associated with IV start procedure today. | Day 0 after completion of the study procedure
  Control subject's assessment of pain level associated with today's IV start procedure:
  Scale 1 - 5; Unable to Evaluate
  1. Not painful at all
  2. Almost no pain
  3. Some pain
  4. Moderate pain
  5. Extreme pain Unable to Evaluate
Subject Satisfaction Survey question for control subject's: Pain associated with today's IV start compared to past IV starts. | Day 0 after completion of the study procedure
  Control subject's assessment of pain associated with today's IV start compared to past IV starts:
  Scale 1 - 5; Unable to Evaluate
  1. Much less pain
  2. Less Painful
  3. Equal Pain
  4. More Painful
  5. Much More Painful Unable to Evaluate
Subject Satisfaction Survey question for control subject's: Anxiety associated with the IV start procedure today. | Day 0 after completion of the study procedure
  Control subject's assessment of anxiety level associated with today's IV start procedure:
  Scale 1 - 5; Unable to Evaluate
  1. Not Anxious
  2. Slightly Anxious
  3. Anxious
  4. Moderately Anxious
  5. Very Anxious Unable to Evaluate
Subject Satisfaction Survey question for control subject's: Anxiety associated with today's IV start compared to past IV starts. | Day 0 after completion of the study procedure
  Control subject's assessment of anxiety level associated with today's IV start procedure compared to past IV starts:
  Scale 1 - 5; Unable to Evaluate
  1. A Lot Less Anxious
  2. Less Anxious
  3. The Same
  4. More Anxious
  5. Very Anxious Unable to Evaluate
Subject Satisfaction Survey question for control subject's: Overall, I was satisfied with today's IV start. | Day 0 after completion of the study procedure
  Control subject's overall assessment of satisfaction with today's IV start:
  Scale 1 - 5; Unable to Evaluate
  1. Strongly Agree
  2. Agree
  3. Neutral
  4. Disagree
  5. Strongly Disagree Unable to Evaluate
Subject Satisfaction Survey question for treatment subject's: Past IV starts have been difficult, uncomfortable or painful. | Day 0 after completion of the study procedure
  Veinplicity subject's assessment of pain associated with past IV starts:
  Scale 1 - 5; Unable to Evaluate
  1. Strongly Agree
  2. Agree
  3. Neutral
  4. Disagree
  5. Strongly Disagree Unable to Evaluate
Subject Satisfaction Survey question for treatment subject's: Today, my IV was started easily. | Day 0 after completion of the study procedure
  Veinplicity subject's assessment of how easy they believe today's IV start was:
  Scale 1 - 5; Unable to Evaluate
  1. Strongly Agree
  2. Agree
  3. Neutral
  4. Disagree
  5. Strongly Disagree Unable to Evaluate
Subject Satisfaction Survey question for treatment subject's: Pain associated with IV start procedure today. | Day 0 after completion of the study procedure
  Veinplicity subject's assessment of pain level associated with today's IV start procedure:
  Scale 1 - 5; Unable to Evaluate
  1. Not painful at all
  2. Almost no pain
  3. Some pain
  4. Moderate pain
  5. Extreme pain Unable to Evaluate
Subject Satisfaction Survey question for treatment subject's: Pain associated with today's IV start compared to past IV starts. | Day 0 after completion of the study procedure
  Veinplicity subject's assessment of pain level associated with today's IV start compared to past IV starts:
  Scale 1 - 5; Unable to Evaluate
  1. Not painful at all
  2. Almost no pain
  3. Some pain
  4. Moderate pain
  5. Extreme pain Unable to Evaluate
Subject Satisfaction Survey question for treatment subject's: Anxiety associated with the IV start procedure today. | Day 0 after completion of the study procedure
  Veinplicity subject's assessment of anxiety level associated with today's IV start procedure:
  Scale 1 - 5; Unable to Evaluate
  1. Not Anxious
  2. Slightly Anxious
  3. Anxious
  4. Moderately Anxious
  5. Very Anxious Unable to Evaluate
Subject Satisfaction Survey question for treatment subject's: Anxiety associated with today's IV start compared to past IV starts. | Day 0 after completion of the study procedure
  Veinplicity subject's assessment of anxiety level associated with today's IV start procedure compared to past IV starts:
  Scale 1 - 5; Unable to Evaluate
  1. A Lot Less Anxious
  2. Less Anxious
  3. The Same
  4. More Anxious
  5. Very Anxious Unable to Evaluate
Subject Satisfaction Survey question for treatment subject's: Pain associated with the Veinplicity stimulation. | Day 0 after completion of the study procedure
  Veinplicity subject's assessment on level of pain associated with today's Veinplicity stimulation:
  Scale 1 - 5; Unable to Evaluate
  1. Not painful at all
  2. Almost no pain
  3. Some pain
  4. Moderate pain
  5. Extreme pain Unable to Evaluate
Subject Satisfaction Survey question for treatment subject's: Veinplicity improved the overall success of my experience. | Day 0 after completion of the study procedure
  Veinplicity subject's assessment on how Veinplicity improved overall success of their experience today:
  1. Strongly Agree
  2. Agree
  3. Neutral
  4. Disagree
  5. Strongly Disagree Unable to Evaluate
Subject Satisfaction Survey question for treatment subject's: The Veinplicity device made it easier for the nurse to find a vein for my IV start today. | Day 0 after completion of the study procedure
  Veinplicity subject's assessment of Veinplicity device made it easier for nurse to find a vein for today's IV start:
  1. Strongly Agree
  2. Agree
  3. Neutral
  4. Disagree
  5. Strongly Disagree Unable to Evaluate
Subject Satisfaction Survey question for treatment subject's: I would choose the Veinplicity again for future IV starts. | Day 0 after completion of the study procedure
  Veinplicity subject's likelihood of choosing to use the Veinplicity device for future IV starts:
  1. Definitely Agree
  2. Agree
  3. Neutral
  4. Disagree
  5. Definitely Disagree Unable to Evaluate
Subject Satisfaction Survey question for treatment subject's: Overall, I was satisfied with today's IV start. | Day 0 after completion of the study procedure
  Veinplicity subject's overall assessment of satisfaction with today's IV start:
  Scale 1 - 5; Unable to Evaluate
  1. Strongly Agree
  2. Agree
  3. Neutral
  4. Disagree
  5. Strongly Disagree Unable to Evaluate
Clinician satisfaction | Assessed on Day 0 after completion of the study procedure
  On Day 0 after each Veinplicity subject's IV procedure, each clinician will complete a Clinician Satisfaction Survey, after cannulation has been attempted and subject is declared either a study success or failure. Clinician's are not to complete this survey for control subjects.
  Scale 1 to 5:
  1. = Strongly Agree
  2. = Moderately Agree
  3. = Neutral
  4. = Moderately Disagree
  5. = Strongly Disagree QUESTION 1: Veinplicity was easy to use. QUESTION 2: Veinplicity improved vein palpability. QUESTION 3: Veinplicity improved vein visualization. QUESTION 4: Veinplicity made it easier to identify a suitable vessel to access.
  QUESTION 5: Veinplicity improved the overall success of the experience. QUESTION 6: Veinplicity resulted in a more positive and less anxious experience for the patient.
  QUESTION 7: I would recommend Veinplicity to a colleague or patient. QUESTION 8: Overall, I was satisfied with using the Veinplicity device.
Change in the vein quality score from baseline to pre-cannulation tourniquet application | Day 0
  scores at baseline and post-stimulation to be assessed at time of tourniquet application by the same clinician.
  Scale = Vessel Health and Preservation (VHP) Peripheral Vein Assessment Scale. Grade 1 = Vein Quality Excellent (4-5 palpable/easily visible veins suitable to cannulate) Grade 2 = Vein Quality Good (2-3 palpable/visible veins suitable to cannulate Grade 3 = Vein Quality Fair (1-2 palpable/visible veins suitable to cannulate [veins may be small, scarred or difficult to find and require heat packs to aid vasodilation]) Grade 4 = Vein Quality Poor (veins not palpable/visible [requires ultrasound assistance or infrared viewer]) Grade 5 = Vein Quality None identifiable (no visible [naked eye or aids] or palpable veins) Fair or Poor indicates to clinician that cannulation may be challenging and require extra time or resources; use of Veinplicity may increase vessel size and improve identification of vessels suitable for cannulation

CONTACTS AND LOCATIONS:
Overall Officials: Gregory J Schears, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Midwest Immunology Clinic and Infusion Center, Plymouth, Minnesota
  - Mayo Clinic-Rochester, Rochester, Minnesota
  - Regions Hospital, Saint Paul, Minnesota